CLINICAL TRIAL: NCT01033643
Title: A Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-3614
Brief Title: A Multiple Dose Study of MK-3614 (MK-3614-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3614-002; MK-3614-002 (Other: Merck); 2009_704 (Other: Merck); 2009-010401-36 (EudraCT Number)
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Results first posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- MK-3614 0.25 mg (Panel A) (Experimental): Participants received 0.25 mg of MK-3614 twice daily (BID) every 12 hours orally for 10 days.
  Interventions: Drug: MK-3614
- MK-3614 0.50/0.25 mg (Panel B) (Experimental): Participants received 0.50 mg of MK-3614 in the morning (AM) and 0.25 mg of MK-3614 in the evening (PM) 12 hours apart orally for 10 days.
  Interventions: Drug: MK-3614
- MK-3614 0.50/0.25 mg (Panel C Repeat) (Experimental): Participants were to receive 0.75 mg of MK-3614 BID every 12 hours orally for 10 Days. Per protocol amendment, the Panel B dose was repeated, and participants received instead 0.50 mg of MK-3614 in the AM, and 0.25 mg of MK-3614 in the PM, 12 hours apart orally for 10 days.
  Interventions: Drug: MK-3614
- MK-3614 0.50 mg (Panel D) (Experimental): Participants received 0.50 mg of MK-3614 three times a day (TID) orally every 8 hours on Day 1 followed by a wash out period for Days 2, 3 and 0.50 mg of MK-3614 every 12 hours orally for 10 days (Days 4-13).
  Interventions: Drug: MK-3614
- MK-3614 0.50 mg (Panel E) (Experimental): Participants were to receive orally 0.50 mg of MK-3614 BID every 12 hours on Day 1 followed by 3 doses (0.50/0.50/0.25 mg) of MK-3614 each 8 hours apart on Day 2; three doses of 0.50 mg of MK-3614 8 hours apart on Days 3,4; and 0.75 mg of MK-3614 BID every 12 hours on Days 5-14. No participants were enrolled in this group.
  Interventions: Drug: MK-3614
- Placebo (All Panels) (Placebo Comparator): Participants received a dose matched placebo orally according to randomization.
  Interventions: Drug: Placebo for MK-3614

INTERVENTIONS:
Drug: MK-3614 — Participants were administered 0.25 mg tablet, orally for a total daily dose according to randomization.
  Arms: MK-3614 0.25 mg (Panel A); MK-3614 0.50 mg (Panel D); MK-3614 0.50 mg (Panel E); MK-3614 0.50/0.25 mg (Panel B); MK-3614 0.50/0.25 mg (Panel C Repeat)
Drug: Placebo for MK-3614 — Participants were administered dose matched placebo tablets according to randomization.
  Arms: Placebo (All Panels)

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple doses of MK-3614 in male participants with mild to moderate hypertension. The primary hypotheses are: 1) Multiple oral doses of MK-3614 are sufficiently safe and well tolerated to permit continued clinical investigation 2) Aortic Augmentation Index (Aix) is reduced 24 hours post the last dose of MK-3614 administered compared to placebo and 3) Increase in the 12-hour weighted averages (TWA 0-12hours) of the heart rate is within 15 beats per minute (bpm) of baseline on first day of multiple dosing of MK-3614 and within 10 bpm of baseline on last day of multiple dosing of MK-3614.

ELIGIBILITY:
Inclusion Criteria:

* Has mild to moderate hypertension
* Has grade 1 or 2 arterial hypertension being treated with a single antihypertensive drug
* Has been a nonsmoker and/or has not used nicotine or nicotine-containing products for at least approximately 6 months; or who have discontinued smoking or the use of nicotine/nicotine-containing products for at least approximately 3 months
* Is in generally good health

Exclusion Criteria:

* Has a history of clinically significant abnormalities or diseases
* Has a history of stroke, chronic seizures, or major neurological disorder
* Has a functional disability that can interfere with rising from a sitting position to the standing position
* Has any personal or family history of a bleeding or a clotting disorder
* Has a history of frequent nose bleeds or has recurrent or active gingivitis
* Has a history of cancer
* Has a history of clinically significant cardiac disease
* Is unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies approximately 2 weeks prior to the administration of study drug
* Consumes excessive amounts of alcohol
* Consumes excessive amounts of caffeinated beverages per day
* Has had major surgery, donated or lost 1 unit of blood or participated in another investigational study within 4 weeks of study
* Has a history of significant multiple and/or severe allergies (including latex) to prescription or non-prescription drugs or food
* Is currently a regular user of any illicit drugs or has a history of drug abuse within approximately 1 year

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-05-27 (Actual); Primary Completion 2009-12-09 (Actual); Study Completion 2009-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 30 participants randomized to the study, received at least one dose of study treatment (All Treated Population) and were evaluable for all safety analysis. No participants were enrolled in Panel E.
Groups:
- MK-3614 0.50/0.25 mg (Panel B): Participants received 0.50 mg of MK-3614 in the morning (AM) and 0.25 mg of MK-3614 in the evening (PM), 12 hours apart orally for 10 days.
- MK-3614 0.50/0.25 mg (Panel C Repeat): Per protocol amendment, the Panel B dose was repeated, and participants received instead 0.50 mg of MK-3614 in the AM, and 0.25 mg of MK-3614 in the PM, 12 hours apart orally for 10 days.
- MK-3614 0.50 mg (Panel D): Participants received single day dose of 0.50 mg of MK-3614 three times a day (TID) every 8 hours on Day 1 followed by a wash out period for Days 2, 3 and multiple doses of 0.50 mg of MK-3614 BID every 12 hours orally for 10 days (Days 4-13).
- MK-3614 0.50 mg (Panel E): Participants were to receive 0.50 mg BID every 12 hours apart or a matching placebo on Day 1 followed by 3 doses (0.50/0.50/0.25 mg) of MK-3614 each 8 hours apart on Day 2, three doses of 0.50 mg of MK-3614 8 hours apart on Days 3, 4 and 0.75 mg of MK-3614 BID every 12 hours on Days 5-14. No participants were enrolled in this group.
Period: Overall Study
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg (Panel D) | MK-3614 0.50 mg (Panel E) | Placebo (All Panels)
Started | 6 | 6 | 6 | 4 | 0 | 8
Completed | 6 | 3 | 6 | 4 | 0 | 7
Not Completed | 0 | 3 | 0 | 0 | 0 | 1
Not completed — Withdrew Consent | 0 | 3 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in Panel E due to study objectives being achieved after enrolling a total of 6 participants (n = 4 received MK-3614; n =2 received placebo) in Panel D.
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg (Panel D) | Placebo (All Panels) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 8 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.7 (5.4) | 48.8 (2.1) | 49.2 (6.1) | 49.3 (8.2) | 45.0 (5.7) | 48.1 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 4 | 8 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 6 | 4 | 8 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 6 | 4 | 8 | 30
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An adverse event was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study intervention, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the study intervention, was also an adverse event. The number of participants who experienced an AE was reported.
Time Frame: Up to approximately 27 days
Population: All participants who received at least one dose of the study treatment. No participants were enrolled in Panel E.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 8
Participants | 4 | 3 | 4 | 3 | 3

2. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An adverse event was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study intervention, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the study intervention, was also an adverse event. The number of participants who discontinued study treatment due to an AE was reported.
Time Frame: Up to approximately 13 days
Population: All participants who received at least one dose of the study treatment. No participants were enrolled in Panel E.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 8
Participants | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Panel A: Area Under the Concentration Time-Curve From 0 to 12 Hours (AUC 0-12hrs) of MK-3614
Description: Blood samples were collected at pre-specified timepoints on first day of multiple dosing of MK-3614 (Day 1) and last day of multiple dosing of MK-3614 (Day 10) to determine the AUC 0-12hrs of MK-3614 in Panel A participants per protocol. AUC 0-12hrs was defined as the area under the concentration-time curve of MK-3614 from time zero to 12 hours postdose.
Time Frame: Days 1, 10: Predose and 1, 2, 4, 6, 8 & 12 hours postdose
Population: All participants in Panel A who received multiple doses of MK-3614, who complied with the protocol sufficiently to ensure that these data exhibited the effects of treatment, according to the underlying scientific model and had available data for the AUC 0-12hrs were evaluated. No participants were enrolled in Panel E.
Measure: Geometric Mean (Standard Deviation); unit: nM*hr
Groups:
- MK-3614 0.50 mg BID (Panel D): Participants received 0.50 mg of MK-3614 BID every 12 hours orally for 10 days (Days 4-13).
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg BID (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 6 | 0 | 0 | 0 | 0
nM*hr
  First Day (Day 1) | 43.9 (8.62) |  |  |  |
  Last Day (Day 10) | 105.0 (24.4) |  |  |  |
Statistical Analysis 1: Comparison: MK-3614 0.25 mg (Panel A); Test type: Other; Accumulation or Geometric Mean Ratio = 2.36 — Accumulation ratio or geometric mean ratio (GMR) was calculated as last day of multiple dosing of MK-3614 (Day 10) divided by the first day of multiple dosing of MK-3614 (Day 1)

4. Primary Outcome: Panel D: Area Under the Concentration Time-Curve From 0 to 12 Hours (AUC 0-12hrs) of MK-3614
Description: Blood samples were collected at pre-specified timepoints to determine the AUC 0-12hrs on first day of multiple dosing of MK-3614 (Day 4) and last day of multiple dosing of MK-3614 (Day 13) to determine the AUC 0-12hrs of MK-3614 in Panel D participants per protocol. AUC 0-12hrs was defined as the area under the concentration-time curve of MK-3614 from time zero to 12 hours postdose.
Time Frame: Days 4, 13: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8 & 12 hours postdose
Population: All participants in Panel D who received multiple doses of MK-3614, who complied with the protocol sufficiently to ensure that these data exhibited the effects of treatment, according to the underlying scientific model and had available data for AUC 0-12hrs were evaluated. No participants were enrolled in Panel E.
Measure: Geometric Mean (Standard Deviation); unit: nM*hr
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg BID (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 0
nM*hr
  First Day (Day 4) |  |  |  | 87.8 (11.0) |
  Last Day (Day 13) |  |  |  | 144.0 (28.1) |
Statistical Analysis 1: Comparison: MK-3614 0.50 mg BID (Panel D); Test type: Other; Accumulation or Geometric Mean Ratio = 1.62 — Accumulation ratio or GMR was calculated as last day of multiple dosing of MK-3614 (Day 13) divided by the first day of multiple dosing of MK-3614 (Day 4)

5. Primary Outcome: Panel D: Area Under the Concentration Time-Curve From 0 to Infinity (AUC 0-inf) of MK-3614
Description: Blood samples were collected at pre-specified timepoints to determine the AUC 0-inf of MK-3614 in Panel D participants who received single daily dosing on Day 1. AUC 0-inf was defined as the area under the concentration-time curve of MK-3614 from time zero to infinity. Geometric mean and 95%CI were not reported because the single day dosing of MK-3614 was only administered on Day 1 for Panel D participants. Instead, AUC 0-24 hours was reported for Panel D participants on Day 1 which is included in the 'other pre-specified outcomes'.
Time Frame: Day 1: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 14, & 24 hours postdose
Population: All participants in Panel D who received single day dose of MK-3614, who complied with the protocol sufficiently to ensure that these data exhibited the effects of treatment, according to the underlying scientific model and had available data for the AUC 0-inf. No participants were enrolled in Panel E.
Groups:
- MK-3614 0.50 mg TID (Panel D): Participants received single day dose of 0.50 mg of MK-3614 three times a day (TID) every 8 hours orally on Day 1.
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg TID (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Panels B, C: Area Under the Concentration Time-Curve From 0 to 24 Hours (AUC 0-24hrs) of MK-3614
Description: Blood samples were collected at pre-specified timepoints to determine the AUC 0-24hrs on first day of multiple dosing of MK-3614 (Day 1) and last day of multiple dosing of MK-3614 (Day 10) to determine the AUC 0-24hrs of MK-3614 in Panel B & C participants per protocol. AUC0-24hrs was defined as the area under the concentration-time curve of MK-3614 from time zero to 24 hours postdose.
Time Frame: Days 1, 10: Predose and 1, 2, 4, 6, 8, 12, 16, & 24 hours postdose
Population: All participants in Panel B & C who received multiple doses of MK-3614, who complied with the protocol sufficiently to ensure that these data exhibited the effects of treatment, according to the underlying scientific model and had available data for AUC 0-24hrs were evaluated. No participants were enrolled in Panel E.
Measure: Geometric Mean (Standard Deviation); unit: nM*hr
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg BID (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 0 | 6 | 6 | 0 | 0
nM*hr
  First Day (Day 1) |  | 188.0 (46.7) | 190.0 (72.3) |  |
  Last Day (Day 10): number analyzed (Participants) | 0 | 3 | 6 | 0 | 0
  Last Day (Day 10) |  | 335.0 (66.1) | 302.0 (82.3) |  |
Statistical Analysis 1: Comparison: MK-3614 0.50/0.25 mg (Panel B); Test type: Other; Accumulation or Geometric Mean Ratio = 1.90 — Accumulation ratio or GMR was calculated as last day of multiple dosing of MK-3614 (Day 10) divided by the first day of multiple dosing of MK-3614 (Day 1)
Statistical Analysis 2: Comparison: MK-3614 0.50/0.25 mg (Panel C Repeat); Test type: Other; Accumulation or Geometric Mean Ratio = 1.63 — [estimate comment as in outcome 6, analysis 1]

7. Primary Outcome: Panel A: Maximum Concentration (Cmax) of MK-3614
Description: Blood samples were collected predose and up to 12 hours postdose on first day of multiple dosing of MK-3614 (Day 1) and last day of multiple dosing (Day 10) for the determination of Cmax in Panel A participants. Cmax was defined as the maximum concentration of MK-3614 reached over 12 hours.
Time Frame: Days 1, 10: Predose and 1, 2, 4, 6, 8 & 12 hours postdose
Population: All participants in Panel A who received multiple doses of MK-3614, who complied with the protocol sufficiently to ensure that these data exhibited the effects of treatment, according to the underlying scientific model and had available data for the Cmax were evaluated. No participants were enrolled in Panel E.
Measure: Geometric Mean (Standard Deviation); unit: nM
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg BID (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 6 | 0 | 0 | 0 | 0
nM
  First Day (Day 1) | 5.61 (1.22) |  |  |  |
  Last Day (Day 10) | 11.6 (2.33) |  |  |  |
Statistical Analysis 1: Comparison: MK-3614 0.25 mg (Panel A); Test type: Other; Accumulation or Geometric Mean Ratio = 1.91 — [estimate comment as in outcome 6, analysis 1]

8. Primary Outcome: Panel D: Maximum Concentration (Cmax) of MK-3614
Description: Blood samples were collected at predose and up to 12 hours postdose on first day of multiple dosing of MK-3614 (Day 4) and last day of multiple dosing of MK-3614 (Day 13) for the determination of Cmax in Panel D participants. Cmax was defined as the maximum concentration of MK-3614 reached over 12 hours after administration of multiple doses of MK-3614.
Time Frame: Days 4, 13: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, & 12 hours postdose
Population: All participants in Panel D who received multiple doses of MK-3614, who complied with the protocol sufficiently to ensure that these data exhibited the effects of treatment, according to the underlying scientific model and had available data for the Cmax were evaluated. No participants were enrolled in Panel E.
Measure: Geometric Mean (Standard Deviation); unit: nM
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg BID (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 0
nM
  First Day (Day 4) |  |  |  | 11.6 (0.85) |
  Last Day (Day 13) |  |  |  | 16.1 (3.04) |
Statistical Analysis 1: Comparison: MK-3614 0.50 mg BID (Panel D); Test type: Other; Accumulation or Geometric Mean Ratio = 1.38 — [estimate comment as in outcome 4, analysis 1]

9. Primary Outcome: Panels B, C: Maximum Concentration (Cmax) of MK-3614
Description: Blood samples were collected at predose and up to 24 hours postdose on first day of multiple dosing of MK-3614 (Day 1) and last day of multiple dosing of MK-3614 (Day 10) for the determination of Cmax in Panel B & C participants. Cmax was defined as the maximum concentration of MK-3614 reached over 24 hours.
Time Frame: Days 1, 10: Predose and 1, 2, 4, 6, 8, 12, 16, & 24 hours postdose
Population: All participants in Panels B, C who received multiple doses of MK-3614, who complied with the protocol sufficiently to ensure that these data exhibited the effects of treatment, according to the underlying scientific model and had available data for the Cmax were evaluated. No participants were enrolled in Panel E.
Measure: Geometric Mean (Standard Deviation); unit: nM
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg BID (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 0 | 6 | 6 | 0 | 0
nM
  First Day (Day 1) |  | 12.2 (1.95) | 11.1 (3.67) |  |
  Last Day (Day 10): number analyzed (Participants) | 0 | 3 | 6 | 0 | 0
  Last Day (Day 10) |  | 19.0 (3.92) | 18.5 (4.92) |  |

10. Primary Outcome: Panel A: Time to Maximum Concentration (Tmax) of MK-3614
Description: Blood samples were collected at predose and up to 12 hours postdose on first day of multiple dosing of MK-3614 (Day 1) and last day of multiple dosing of MK-3614 (Day 10) to determine the Tmax in Panel A participants. Tmax was defined as time to the maximum concentration of MK-3614 reached over 12 hours.
Time Frame: Days 1, 10: Predose and 1, 2, 4, 6, 8, & 12 hours postdose
Population: All participants in Panel A who received multiple doses of MK-3614, who complied with the protocol sufficiently to ensure that these data exhibited the effects of treatment, according to the underlying scientific model and had available data for the Tmax were evaluated. No participants were enrolled in Panel E.
Measure: Median (Full Range); unit: hr
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg BID (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 6 | 0 | 0 | 0 | 0
hr
  First Day (Day 1) | 4.0 [4.0 to 6.0] |  |  |  |
  Last Day (Day 10) | 4.0 [2.0 to 4.0] |  |  |  |

11. Primary Outcome: Panel D: Time to Maximum Concentration (Tmax) of MK-3614
Description: Blood samples were collected at predose and up to 12 hours on first day of multiple dosing of MK-3614 (Day 4) and last day of multiple dosing of MK-3614 (Day 13) to determine the Tmax in Panel D participants. Tmax was defined as time to the maximum concentration of MK-3614 reached over 12 hours among participants in Panel D.
Time Frame: Days 4, 13: Predose and 0.5, 1, 2, 3 ,4, 5, 6, 8 & 12 hours postdose
Population: All participants in Panel D who received multiple doses of MK-3614, who complied with the protocol sufficiently to ensure that these data exhibited the effects of treatment, according to the underlying scientific model and had available data for the Tmax. No participants were enrolled in Panel E.
Measure: Median (Full Range); unit: hr
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg BID (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 0
hr
  First Day (Day 4) |  |  |  | 4.5 [4.0 to 5.0] |
  Last Day (Day 13) |  |  |  | 4.5 [3.0 to 5.0] |

12. Primary Outcome: Panels B, C: Time to Maximum Concentration (Tmax) of MK-3614
Description: Blood samples were collected at predose and up to 24 hours on first day of multiple dosing of MK-3614 (Day 1) and last day of multiple dosing of MK-3614 (Day 10) to determine the Tmax in Panel B & C participants. Tmax was defined as time to the maximum concentration of MK-3614 reached over 24 hours.
Time Frame: Days 1, 10: Predose and 1, 2, 4, 6, 8, 12, 16, & 24 hours postdose
Population: All participants in Panels B & C who received multiple doses of MK-3614, who complied with the protocol sufficiently to ensure that these data exhibited the effects of treatment, according to the underlying scientific model and had available data for the Tmax were evaluated. No participants were enrolled in Panel E.
Measure: Median (Full Range); unit: hr
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg BID (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 0 | 6 | 6 | 0 | 0
hr
  First Day (Day 1) |  | 4.0 [4.0 to 24.0] | 11.0 [4.0 to 24.0] |  |
  Last Day (Day 10): number analyzed (Participants) | 0 | 3 | 6 | 0 | 0
  Last Day (Day 10) |  | 6.0 [4.0 to 6.0] | 4.0 [4.0 to 6.0] |  |

13. Primary Outcome: Panels A, B & C: Apparent Terminal Half-Life (t1/2) of MK-3614
Description: Blood samples were collected at pre-specified time points on Day 10 to determine t½ in Panels A, B, & C participants who received multiple doses of MK-3614. Apparent t½ was defined as the time required to eliminate half the amount of MK-3614 from plasma concentration.
Time Frame: Day 10: Predose and 1, 2, 4, 6, 8, 12, 16, 24, 36, & 48 hours postdose
Population: All participants in Panels A, B, & C who received multiple doses of MK-3614, who complied with the protocol sufficiently to ensure that these data exhibited the effects of treatment, according to the underlying scientific model and had available data for the t1/2 were evaluated. No participants were enrolled in Panel E.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg BID (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 6 | 3 | 6 | 0 | 0
hr | 10.1 (0.7) | 12.7 (1.2) | 11.9 (2.7) |  |

14. Primary Outcome: Panel D: Apparent Terminal Half-Life (t1/2) of MK-3614
Description: Blood samples were collected at pre-specified time points on Day 13 to determine t½ in Panel D participants who received multiple doses of MK-3614. Apparent t½ was defined as the time required to eliminate half the amount of MK-3614 from plasma concentration.
Time Frame: Day 13: Predose and 0.5 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, & 48 hours postdose
Population: All participants in Panel D who received multiple doses of MK-3614, who complied with the protocol sufficiently to ensure that these data exhibited the effects of treatment, according to the underlying scientific model and had available data for the t1/2 were evaluated. No participants were enrolled in Panel E.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg BID (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 0
hr |  |  |  | 8.1 (1.3) |

15. Primary Outcome: Change From Baseline in Aortic Augmentation Index (AIx) at 24 Hours Postdose After Multiple Doses of MK-3614 or Placebo
Description: Aortic AIx is the percentage of the central pulse pressure attributed to the reflected pulse wave, and is an indirect measure of systemic arterial stiffness. Aortic AIx was measured at pre-specified timepoints by aplanation tonometry of radial artery. Linear model containing panel as a fixed effect was used to report the change from baseline in aortic Aix at 24 hours postdose. The 90% confidence intervals (CIs) for the true mean difference (MK-3614-placebo) in change from baseline were obtained using the mean square error from the linear model. Placebo data was pooled across all panels for the analysis. A decrease in the point estimate of ≥ 5 percentage points was considered clinically meaningful.
Time Frame: Panels A, B & C: Day 10: Baseline & 24 hours postdose; Panel D: Day 13: Baseline & 24 hours postdose; Placebo: Day 10 or Day 13: Baseline & 24 hours postdose
Population: All participants who received multiple doses of MK-3614 or a matching placebo, who complied with the protocol sufficiently to ensure that these data exhibited the effects of treatment, according to the underlying scientific model and had a baseline and at least one post baseline AIx value available on last day (Day 10 for Panels A, B, C and Day 13 on Panel D) were evaluated. No participants were enrolled in Panel E.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage of central pulse pressure
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg BID (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 6 | 3 | 6 | 4 | 7
Percentage of central pulse pressure | -9.94 [-14.32 to -5.57] | -1.0 [-6.36 to 4.36] | -9.25 [-13.04 to -5.46] | -2.25 [-6.04 to 1.54] | -5.78 [-8.87 to -2.68]
Statistical Analysis 1: Comparison: MK-3614 0.25 mg (Panel A) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = -4.17, 90% CI 2-sided [-9.53 to 1.20]
Statistical Analysis 2: Comparison: MK-3614 0.50/0.25 mg (Panel B) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = 4.78, 90% CI 2-sided [-1.41 to 10.97]
Statistical Analysis 3: Comparison: MK-3614 0.50/0.25 mg (Panel C Repeat) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = -3.47, 90% CI 2-sided [-8.37 to 1.42]
Statistical Analysis 4: Comparison: MK-3614 0.50 mg BID (Panel D) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = 3.53, 90% CI 2-sided [-1.37 to 8.42]

16. Secondary Outcome: Change From Baseline in Time-Weighted Average Across 12 Hours (TWA 0-12hrs) of Peripheral Systolic Blood Pressure (SBP) on First Day of Multiple Dosing of MK-3614 or Placebo
Description: Peripheral SBP was measured by the SphygmoCor® device. TWA 0-12hrs was obtained as follows: For all peripheral SBP values obtained over the 12-hour observation period (1, 2, 3, 4, 5, 6, 8, 10, 12 hours postdose), multiplied the length of time that the participant spent at each peripheral SBP value by that peripheral SBP value, added these products together, and then divided by duration of the observation period. Multiple dose effects of MK-3614 or placebo on peripheral SBP were estimated as a TWA change from baseline (0 hours) over the 12 hour postdose on first day of multiple dosing (Panels A, B, C: Day 1; Panel D: Day 4) and summarized descriptively. Placebo data was pooled across all panels for the analysis. Linear model containing panel as a fixed effect was used report the mean difference from placebo and associated 90% CIs after multiple doses of MK-3614 or placebo.
Time Frame: Panels A, B, C: Day 1: Baseline (0 hours) & up to 12 hours postdose; Panel D: Day 4: Baseline (0 hours) & up to 12 hours postdose; Placebo: Day 1 or Day 4: Baseline (0 hours) & up to 12 hours postdose
Population: All participants who received multiple doses of MK-3614 or a matching placebo, who complied with the protocol sufficiently to ensure that these data exhibited the effects of treatment, according to the underlying scientific model and had available data for the SBP were evaluated. No participants were enrolled in Panel E.
Measure: Mean (Full Range); unit: mm Hg
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg BID (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 8
mm Hg | -9.47 [-26.08 to 3.69] | -15.19 [-26.61 to -7.83] | -14.36 [-31.53 to -6.29] | -5.57 [-8.88 to 1.06] | -5.88 [-26.60 to 7.01]
Statistical Analysis 1: Comparison: MK-3614 0.25 mg (Panel A) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = 0.23, 90% CI 2-sided [-6.91 to 7.36]
Statistical Analysis 2: Comparison: MK-3614 0.50/0.25 mg (Panel B) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = -1.66, 90% CI 2-sided [-8.79 to 5.47]
Statistical Analysis 3: Comparison: MK-3614 0.50/0.25 mg (Panel C Repeat) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = 2.11, 90% CI 2-sided [-5.02 to 9.25]
Statistical Analysis 4: Comparison: MK-3614 0.50 mg BID (Panel D) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = -1.23, 90% CI 2-sided [-9.41 to 6.94]

17. Secondary Outcome: Change From Baseline in Time-Weighted Average Across 12 Hours (TWA 0-12hrs) of Peripheral Systolic Blood Pressure (SBP) on Last Day After Multiple Dosing of MK-3614 or Placebo
Description: Peripheral SBP was measured by the SphygmoCor® device. TWA 0-12hrs was obtained as follows: For all peripheral SBP values obtained over the 12-hour observation period (1, 2, 3, 4, 5, 6, 8, 10, and 12 hours postdose), multiplied the length of time that the participant spent at each peripheral SBP value by that peripheral SBP value, added these products together, and then divided by duration of the observation period. Multiple dose effects of MK-3614 or placebo on peripheral SBP were estimated as a TWA change from baseline (0 hours) over the 12 hour postdose on last day of multiple dosing (Panels A, B, C: Day 10; Panel D: Day 13) and summarized descriptively. Placebo data was pooled across all panels for the analysis. Linear model containing panel as a fixed effect was used report the mean difference from placebo and associated 90% CIs after multiple doses of MK-3614 or placebo.
Time Frame: Panels A, B, C: Day 1: Baseline (0 hours) & up to 12 hours; Panel D: Day 4: Baseline (0 hours) & up to 12 hours; Placebo: Day 1 or Day 4: Baseline (0 hours) & up to 12 hours
Population: as for outcome 16
Measure: Mean (Full Range); unit: mm Hg
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg BID (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 6 | 3 | 6 | 4 | 7
mm Hg | -10.25 [-32.22 to 3.89] | -19.33 [-28.50 to -11.82] | -15.61 [-38.92 to -0.01] | -14.05 [-19.54 to -6.81] | -8.29 [-20.51 to 0.85]
Statistical Analysis 1: Comparison: MK-3614 0.25 mg (Panel A) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = -0.75, 90% CI 2-sided [-9.29 to 7.79]
Statistical Analysis 2: Comparison: MK-3614 0.50/0.25 mg (Panel B) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = -3.73, 90% CI 2-sided [-14.32 to 6.86]
Statistical Analysis 3: Comparison: MK-3614 0.50/0.25 mg (Panel C Repeat) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = 0.66, 90% CI 2-sided [-7.88 to 9.20]
Statistical Analysis 4: Comparison: MK-3614 0.50 mg BID (Panel D) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = -9.92, 90% CI 2-sided [-19.54 to -0.30]

18. Secondary Outcome: Change From Baseline in Time-Weighted Average Across 24 Hours (TWA 0-24hrs) of Peripheral Systolic Blood Pressure (SBP) on Last Day of Multiple Dosing of MK-3614 or Placebo
Description: Peripheral SBP was measured by the SphygmoCor® device. TWA 0-24hrs was obtained as follows: For all peripheral SBP values obtained over the 24-hour observation period (1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, and 24 hours postdose), multiplied the length of time that the participant spent at each peripheral SBP value by that peripheral SBP value, added these products together, and then divided by duration of the observation period. Multiple dose effects of MK-3614 or placebo on peripheral SBP were estimated as a TWA change from baseline (0 hours) over the 24 hour postdose on last day of multiple dosing (Panels A, B & C - Day 10; Panel D - Day 13) and summarized descriptively. Placebo data was pooled across all panels for the analysis. Linear model containing panel as a fixed effect was used report the mean difference from placebo and associated 90% CIs after multiple doses of MK-3614 or placebo.
Time Frame: Panels A, B, C: Day 10: Baseline (0 hours) & up to 24 hours postdose; Panel D: Day 13: Baseline (0 hours) & up to 24 hours postdose; Placebo: Day 10 or Day 13: Baseline (0 hours) & up to 24 hours postdose
Population: as for outcome 16
Measure: Mean (Full Range); unit: mm Hg
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg BID (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 6 | 3 | 6 | 4 | 7
mm Hg | -11.37 [-34.75 to 6.58] | -18.59 [-27.29 to -11.51] | -17.66 [-42.57 to -5.52] | -15.43 [-18.42 to -7.11] | -9.15 [-20.30 to -2.03]
Statistical Analysis 1: Comparison: MK-3614 0.25 mg (Panel A) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = -1.02, 90% CI 2-sided [-9.36 to 7.32]
Statistical Analysis 2: Comparison: MK-3614 0.50/0.25 mg (Panel B) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = -2.12, 90% CI 2-sided [-12.47 to 8.22]
Statistical Analysis 3: Comparison: MK-3614 0.50/0.25 mg (Panel C Repeat) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = -0.53, 90% CI 2-sided [-8.87 to 7.81]
Statistical Analysis 4: Comparison: MK-3614 0.50 mg BID (Panel D) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = -10.44, 90% CI 2-sided [-19.83 to -1.04]

19. Secondary Outcome: Change From Baseline in Time-Weighted Average Across 12 Hours (TWA 0-12hrs) of Peripheral Diastolic Blood Pressure (DBP) on First Day of Multiple Dosing of MK-3614 or Placebo
Description: Peripheral DBP was measured by the SphygmoCor® device. TWA 0-12hrs was obtained as follows: For all peripheral DBP values obtained over the 12-hour observation period (1, 2, 3, 4, 5, 6, 8, 10, and 12 hours postdose), multiplied the length of time that the participant spent at each peripheral DBP value by that peripheral DBP value, added these products together, and then divided by duration of the observation period. Multiple dose effects of MK-3614 or placebo on peripheral DBP were estimated as a TWA change from baseline (0 hours) over the 12 hour postdose on first day of multiple dosing (Panels A, B, C: Day 1; Panel D: Day 4) and summarized descriptively. Placebo data was pooled across all panels for the analysis. Linear model containing panel as a fixed effect was used report the mean difference from placebo and associated 90% CIs after multiple doses of MK-3614 or placebo.
Time Frame: as for outcome 16
Population: All participants who received multiple doses of MK-3614 or a matching placebo, who complied with the protocol sufficiently to ensure that these data exhibited the effects of treatment, according to the underlying scientific model and had available data for the DBP were evaluated. No participants were enrolled in Panel E.
Measure: Mean (Full Range); unit: mm Hg
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg BID (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 8
mm Hg | -8.32 [-16.63 to -1.82] | -13.18 [-21.01 to -5.75] | -9.85 [-18.72 to -2.92] | -3.97 [-9.51 to 0.85] | -3.17 [-9.64 to 4.51]
Statistical Analysis 1: Comparison: MK-3614 0.25 mg (Panel A) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = -1.73, 90% CI 2-sided [-6.50 to 3.04]
Statistical Analysis 2: Comparison: MK-3614 0.50/0.25 mg (Panel B) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = -4.23, 90% CI 2-sided [-9.00 to 0.54]
Statistical Analysis 3: Comparison: MK-3614 0.50/0.25 mg (Panel C Repeat) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = -1.05, 90% CI 2-sided [-5.82 to 3.72]
Statistical Analysis 4: Comparison: MK-3614 0.50 mg BID (Panel D) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = -2.00, 90% CI 2-sided [-3.46 to 7.46]

20. Secondary Outcome: Change From Baseline in Time-Weighted Average Across 12 Hours (TWA 0-12hrs) of Peripheral Diastolic Blood Pressure (DBP) on Last Day of Multiple Dosing of MK-3614 or Placebo
Description: Peripheral DBP was measured by the SphygmoCor® device. TWA 0-12hrs was obtained as follows: For all peripheral DBP values obtained over the 12-hour observation period (1, 2, 3, 4, 5, 6, 8, 10, and 12 hours postdose), multiplied the length of time that the participant spent at each peripheral DBP value by that peripheral DBP value, added these products together, and then divided by duration of the observation period. Multiple dose effects of MK-3614 or placebo on peripheral DBP were estimated as a TWA change from baseline (0 hours) over the 12 hour postdose on last day of multiple dosing (Panels A, B, C: Day 10; Panel D: Day 13) and summarized descriptively. Placebo data was pooled across all panels for the analysis. Linear model containing panel as a fixed effect was used report the mean difference from placebo and associated 90% CIs after multiple doses of MK-3614 or placebo.
Time Frame: Panels A, B, C: Day 10: Baseline (0 hours) & up to 12 hours postdose; Panel D: Day 13: Baseline (0 hours) & up to 12 hours postdose; Placebo: Day 10 or Day 13: Baseline (0 hours) & up to 12 hours postdose
Population: All participants who received multiple doses of MK-3614 or a matching placebo, who received multiple doses of MK-3614, who complied with the protocol sufficiently to ensure that these data exhibited the effects of treatment, according to the underlying scientific model and had available data for the DBP were evaluated. No participants were enrolled in Panel E.
Measure: Mean (Full Range); unit: mm Hg
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg BID (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 6 | 3 | 6 | 4 | 7
mm Hg | -10.81 [-21.67 to -3.29] | -15.43 [-24.79 to -10.50] | -10.50 [-22.11 to -2.21] | -8.58 [-14.51 to -3.78] | -3.43 [-9.74 to 8.40]
Statistical Analysis 1: Comparison: MK-3614 0.25 mg (Panel A) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = -3.87, 90% CI 2-sided [-9.37 to 1.64]
Statistical Analysis 2: Comparison: MK-3614 0.50/0.25 mg (Panel B) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = -7.20, 90% CI 2-sided [-14.03 to -0.37]
Statistical Analysis 3: Comparison: MK-3614 0.50/0.25 mg (Panel C Repeat) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = -1.33, 90% CI 2-sided [-6.83 to 4.18]
Statistical Analysis 4: Comparison: MK-3614 0.50 mg BID (Panel D) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = -2.24, 90% CI 2-sided [-8.45 to 3.96]

21. Secondary Outcome: Change From Baseline in Time-Weighted Average Across 24 Hours (TWA 0-24hrs) of Peripheral Diastolic Blood Pressure (DBP) on Last Day of Multiple Dosing of MK-3614 or Placebo
Description: Peripheral DBP was measured by the SphygmoCor® device. TWA 0-24hrs was obtained as follows: For all peripheral DBP values obtained over the 24-hour observation period (1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, and 24 hours postdose), multiplied the length of time that the participant spent at each peripheral DBP value by that peripheral DBP value, added these products together, and then divided by duration of the observation period. Multiple dose effects of MK-3614 or placebo on peripheral DBP were estimated as a TWA change from baseline (0 hours) over the 12 hour postdose on last day of multiple dosing (Panels A, B, C: Day 10; Panel D: Day 13) and summarized descriptively. Placebo data was pooled across all panels for the analysis. Linear model containing panel as a fixed effect was used report the mean difference from placebo and associated 90% CIs after multiple doses of MK-3614 or placebo.
Time Frame: as for outcome 18
Population: as for outcome 20
Measure: Mean (Full Range); unit: mm Hg
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg BID (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 6 | 3 | 6 | 4 | 7
mm Hg | -10.43 [-22.92 to -2.12] | -15.64 [-23.27 to -11.54] | -10.65 [-22.06 to -6.24] | -9.89 [-14.24 to -5.03] | -4.17 [-10.94 to 7.85]
Statistical Analysis 1: Comparison: MK-3614 0.25 mg (Panel A) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = -2.74, 90% CI 2-sided [-7.92 to 2.43]
Statistical Analysis 2: Comparison: MK-3614 0.50/0.25 mg (Panel B) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = -6.67, 90% CI 2-sided [-13.09 to -0.25]
Statistical Analysis 3: Comparison: MK-3614 0.50/0.25 mg (Panel C Repeat) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = -0.74, 90% CI 2-sided [-5.91 to 4.44]
Statistical Analysis 4: Comparison: MK-3614 0.50 mg BID (Panel D) vs Placebo (All Panels); Test type: Other — Linear Model; Mean Difference from Placebo = -2.81, 90% CI 2-sided [-8.64 to 3.02]

22. Secondary Outcome: Panels B, C, & D: Change From Baseline in Bleeding Time (BT) at 5 Hours Postdose on Last Day After Multiple Doses of MK-3614 or Placebo
Description: Blood was drawn at baseline (0 hours) and 5 hours postdose on last day (Panels B, C: Day 10; Panel D: Day 13 per protocol) to assess bleeding time using a Newborn Surgicutt device. Linear model containing panel as a fixed effect was used to generate fold change from baseline and associated 90% CIs. Placebo data was pooled across panels B, C and D for the analysis.
Time Frame: Panels B, C: Day 10: Baseline (0 hours) & 5 hours postdose; Panel D: Day 13: Baseline (0 hours) & 5 hours postdose; Placebo: Day 10 or Day 13: Baseline (0 hours) & 5 hours postdose
Population: All participants in Panels B, C & D who received multiple doses of MK-3614 or a matching placebo, who complied with the protocol sufficiently to ensure that these data exhibited the effects of treatment, according to the underlying scientific model and had available data for the BT were evaluated. No participants were enrolled in Panel E.
Measure: Least Squares Mean (90% Confidence Interval); unit: seconds
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg BID (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 0 | 3 | 6 | 4 | 5
seconds |  | 1.21 [0.70 to 2.08] | 0.61 [0.40 to 0.94] | 1.23 [0.77 to 1.97] | 1.29 [0.85 to 1.96]
Statistical Analysis 1: Comparison: MK-3614 0.50/0.25 mg (Panel B) vs Placebo (All Panels); Test type: Other — Linear Model; Geometric Mean Ratio (GMR) = 0.94, 90% CI 2-sided [0.47 to 1.87] — GMR was calculated as MK-3614 Dose divided by Placebo
Statistical Analysis 2: Comparison: MK-3614 0.50/0.25 mg (Panel C Repeat) vs Placebo (All Panels); Test type: Other — Linear Model; Geometric Mean Ratio (GMR) = 0.48, 90% CI 2-sided [0.26 to 0.87] — GMR was calculated as MK-3614 Dose divided by Placebo
Statistical Analysis 3: Comparison: MK-3614 0.50 mg BID (Panel D) vs Placebo (All Panels); Test type: Other — Linear Model; Geometric Mean Ratio (GMR) = 0.95, 90% CI 2-sided [0.51 to 1.79] — GMR was calculated as MK-3614 Dose divided by Placebo

23. Secondary Outcome: Cyclic Guanosine Monophosphate (cGMP) Concentration Levels After Multiple Doses of MK-3614
Description: Whole Blood was drawn at predose (baseline) and at 4, 24 hours postdose on last day of multiple dosing of MK-3614 (Panels A, B & C: Day 10; Panel D: Day 13) to measure cGMP concentration levels. Linear mixed effects model containing panel, time, and panel by time interaction as fixed effects and participant within panel as a random effect was used to generate geometric mean and associated 90% CIs. Placebo data was pooled across all panels for the analysis.
Time Frame: Panels A, B & C: Day 10: Predose & 4, 24 hours postdose; Panel D: Day 13: Predose & 4, 24 hours postdose; Placebo: Day 10 or Day 13: Predose & 4, 24 hours postdose
Population: All participants who received multiple doses of MK-3614 or a matching placebo, who complied with the protocol sufficiently to ensure that these data exhibited the effects of treatment, according to the underlying scientific model and had available data for the cGMP. No participants were enrolled in Panel E.
Measure: Geometric Mean (90% Confidence Interval); unit: pmole cGMP/g protein
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg BID (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 6 | 3 | 6 | 4 | 7
pmole cGMP/g protein
  Predose | 443.55 [327.44 to 600.82] | 507.86 [330.63 to 780.00] | 517.34 [381.95 to 700.78] | 405.57 [279.7 to 588.16] | 269.72 [203.65 to 357.20]
  4 Hours | 515.43 [380.51 to 698.13] | 532.62 [346.78 to 818.11] | 721.33 [532.51 to 977.01] | 394.89 [272.30 to 572.66] | 316.43 [233.62 to 428.63]
  24 Hours | 456.28 [336.84 to 618.07] | 627.72 [408.71 to 964.20] | 567.14 [418.68 to 768.16] | 497.20 [342.85 to 721.04] | 262.41 [198.13 to 347.51]

24. Other Pre Specified Outcome: Panel D: Area Under the Concentration Time-Curve From Hour 0 to 24 Hours (AUC 0-24hrs) of MK-3614
Description: Blood samples were collected at pre-specified timepoints to determine the AUC 0-24hrs of MK-3614 in Panel D participants who received single daily dosing on Day 1. AUC 0-24hrs was defined as the area under the concentration-time curve of MK-3614 from time zero to 24 hours. AUC 0-24hrs was reported instead of AUC 0-inf since Panel D participants received single daily dosing only on Day 1.
Time Frame: Day 1: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 14, & 24 hours postdose
Population: All participants in Panel D who received single day dose of MK-3614, who complied with the protocol sufficiently to ensure that these data exhibited the effects of treatment, according to the underlying scientific model and had available data for the AUC 0-24 hours were evaluated. No participants were enrolled in Panel E.
Measure: Geometric Mean (Standard Deviation); unit: nM*hr
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg TID (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 0
nM*hr |  |  |  | 290.0 (39.6) |

25. Primary Outcome: Time-weighted Average Across 12 Hours (TWA 0-12hrs) for Heart Rate (HR) After Administration of MK-3614 or Placebo
Description: HR was measured with a validated automatic device. TWA 0-12hrs equals all HR values over 12-hr observation period multiplied by length of time participant spent at each HR value by that HR value; added products together,& divided by observation period duration. Linear mixed effects model with panel, day, panel by day interaction as fixed effects & participant-within-panel as random effect was used to generate TWA 0-12hrs on 1st day of single dosing (Panel D: Day 1) or 1st day of multiple dosing of MK-3614/placebo (Panels A,B,C: Day 1; Panel D: Day 4) and last day of multiple dosing of MK-3614/placebo (Panels A,B,C: Day 10; Panel D: Day 13) & 90% CIs for true TWA using appropriate components of variance. Pooled placebo data at Day 1 indicates first day of single dosing (Panel D: Day 1) & first day of multiple dosing of placebo (Panels A,B,C: Day 1; Panel D: Day 4) & at Day 10 indicates last day of multiple dosing of placebo from all panels (Panels A,B,C: Day 10; Panel D: Day 13).
Time Frame: Panels A, B, C: Days 1, 10: Predose & 1, 2, 3, 4, 5, 6, 8, 10, 12 hours postdose; Panel D: Days 1, 4, 13: Predose & 1, 2, 3, 4, 5, 6, 8, 10, 12 hours postdose; Placebo: Days 1 & 10 or 1, 4, 13: Predose & 1, 2, 3, 4, 5, 6, 8, 10, 12 hours postdose
Population: All participants who received MK-3614 dose or a matching placebo, who complied with the protocol sufficiently to ensure that these data exhibited the effects of treatment, according to the underlying scientific model and had available data for the HR were evaluated. Due to differing dosing schedules, some time points were not applicable for certain arms (indicated by zero participants analyzed entered in the table). No participants were enrolled in Panel E.
Measure: Least Squares Mean (90% Confidence Interval); unit: beats per minute (bpm)
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg (Panel D) | Placebo (All Panels)
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 8
beats per minute (bpm)
  Day 1 | 62.15 [60.92 to 63.37] | 63.58 [62.36 to 64.80] | 63.04 [61.82 to 64.27] | 69.84 [68.26 to 71.42] | 66.80 [65.84 to 67.76]
  Day 4: number analyzed (Participants) | 0 | 0 | 0 | 4 | 0
  Day 4 |  |  |  | 70.18 [66.68 to 71.67] |
  Day 10: number analyzed (Participants) | 6 | 3 | 6 | 0 | 7
  Day 10 | 61.12 [59.90 to 62.34] | 63.00 [61.28 to 64.73] | 65.61 [64.39 to 66.83] |  | 66.76 [65.63 to 67.89]
  Day 13: number analyzed (Participants) | 0 | 0 | 0 | 4 | 0
  Day 13 |  |  |  | 69.82 [68.32 to 71.32] |

ADVERSE EVENTS:
Time Frame: Non-serious AEs, serious AEs and all-cause mortality were collected for up to approximately 27 days.
Description: All-Cause mortality is reported for all enrolled participants. Serious AEs and Other AEs were reported for all randomized participants who received at least 1 dose of study treatment. No participants were enrolled in Panel E since the study objectives were achieved after enrolling 4 participants in Panel D.
Arm/Group | MK-3614 0.25 mg (Panel A) | MK-3614 0.50/0.25 mg (Panel B) | MK-3614 0.50/0.25 mg (Panel C Repeat) | MK-3614 0.50 mg (Panel D) | Placebo (All Panels)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/4 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/4 | 0/8
Other Adverse Events (participants affected / at risk) | 4/6 | 3/6 | 4/6 | 3/4 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-3614 0.25 mg (Panel A) (N=6) | MK-3614 0.50/0.25 mg (Panel B) (N=6) | MK-3614 0.50/0.25 mg (Panel C Repeat) (N=6) | MK-3614 0.50 mg (Panel D) (N=4) | Placebo (All Panels) (N=8)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces pale (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (3) | 1 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Peripheral paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Visual field defect (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.